CLINICAL TRIAL: NCT05508516
Title: The Efficacy and Safety of the Shugan Dingtong Decoction in the Treatment of Fibromyalgia
Brief Title: Shugan Dingtong Decoction in the Treatment of Fibromyalgia
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Yuan Xu, professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LZhang
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Shugan Dingtong decoction (Experimental): Patients will accept Shugan Dingtong decoction 150ml (twice, per day) for 12 weeks.
  Interventions: Drug: Shugan Dingtong decoction
- duloxetine hydrochloride (Active Comparator): Patients will accept duloxetine hydrochloride 20mg (twice, per day) for 12 weeks.
  Interventions: Drug: Duloxetine Hydrochloride

INTERVENTIONS:
Drug: Shugan Dingtong decoction — Patients will accept Shugan Dingtong decoction 150ml (twice, per day) for 12 weeks.
  Arms: Shugan Dingtong decoction
Drug: Duloxetine Hydrochloride — Patients will accept duloxetine hydrochloride 20mg (twice, per day) for 12 weeks.
  Arms: duloxetine hydrochloride

SUMMARY:
Fibromyalgia (FM) is a syndrome characterized by chronic and widespread musculoskeletal pain, fatigue sleep disturbances and cognitive and somatic symptoms. It is commonly conjectured that central sensitization is physiological hallmark of FM. Therefore, centrally acting medications including antidepressants and anticonvulsants are used to treat FM via downregulating dorsal horn sensitization and systemic hyperexcitability.However, those drugs are limited in clinical practice resulting from dose-limiting adverse effects and incomplete drug efficacy.Shugan Dingtong decoction(SGDTD) is a Chinese herbal formula and has been used for treatment of FM in clinical practice many years. However, few research can provide high-quality evidence on the efficacy and safety of SGDTD for the treatment of FM. Therefore, a parallel-group randomized controlled trial was designed to evaluate the efficacy and safety of SGDTD on FM.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-70 years old.
* patients who meet the diagnostic criteria of American College of Rheumatology in 2016.
* patients who meet the diagnostic criteria of Syndrome of stagnation of liver qi.
* pain scores between3 and 7 on visual analogue scale.
* patients sign the informed consent forms.

Exclusion Criteria:

* pregnant and lactating women.
* patients with serious primary diseases of respiratory, digestive, urinary, cardiovascular and immune system.
* patients with mental and psychological disorders including cognitive im-pairment, severe depression, somatoform disorders.
* patients with secondary fibromyalgia resulted from osteoarthritis, rheumatoid arthritis, trauma, hypothyroidism, malignant tumor.
* patients with severe pain resulted from diabetic and postherpetic neuralgia.
* patients who are allergic to the drugs used in this study.
* patients are participation in any other clinical trials or receive other drugs for the treatment of fibromyalgia.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2024-10-18 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale pain scores | 12 Weeks
  The primary outcome of this study is visual analogue scale(VAS) pain score used to evalu-ate pain intensity. VAS pain score ranges from 0 to 10, where 0 refers to no pain and 10 refers to unbearable pain.

SECONDARY OUTCOMES:
Fibromyalgia impact questionnaire | 12 Weeks
  The fibromyalgia impact questionnaire will be used to measure physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well being. This score ranges from 0 to 100 and high scores are related to greater impact on life quality.
Fatigue scale-14 | 12 Weeks
  The fatigue scale-14 will be used to evaluate physical and mental fatigue. The higher the score, the greater the fatigue.
Pittsburgh sleep quality index | 12 Weeks
  Pittsburgh sleep quality index will be used to assess the sleep quality within the past month. The higher the score, the worse sleep quality. A total of PSQI score greater than five yielded a diagnostic sensitivity of 89.6% and specificity of 86.5%
Traditional Chinses medicine symptom score | 12 Weeks
  Traditional Chinses medicine symptom score is calculated based on the percentage of symptom score reduction

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Lan T, Zhang Y, Guo Z, Yu H, Sun G, Wang Z, Yan Z, Tao Q, Xu Y. Osteoarthritis and Degree of Fatigue are Associated with Pain Levels in Patients with Fibromyalgia Syndrome: A Cross-Sectional Study of 394 Patients. Int J Gen Med. 2025 Jan 31;18:497-507. doi: 10.2147/IJGM.S503902. eCollection 2025. PMID 39906173